CLINICAL TRIAL: NCT07298525
Title: Safety Exploration and Evaluation of Dexmedetomidine Hydrochloride Nasal Spray for Pre-anesthesia Sedation in Low-Monitoring Settings
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Li, Chief Physician, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPPH2025586
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dexmedetomidine; Sedation; Safety; Preanesthetic Medication; Monitored Anaesthesia Care
Keywords: Dexmedetomidine; Sedation; Safety; Preanesthetic Medication; Monitored Anaesthesia Care; Adverse Events of Respiratory Circulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1(LD): Dexmedetomidine hydrochloride nasal spray 50μg, and placebo nasal spray 50μg (Experimental)
  Interventions: Drug: Dexmedetomidine hydrochloride nasal spray
- Group 2(HD): Dexmedetomidine hydrochloride nasal spray 100μg (Experimental)
  Interventions: Drug: Dexmedetomidine hydrochloride nasal spray
- Group 3(C): Placebo nasal spray 100μg (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine hydrochloride nasal spray — Group 1 (LD) was administered 50 μg of dexmedetomidine hydrochloride nasal spray and 50 μg of placebo nasal spray
  Arms: Group 1(LD): Dexmedetomidine hydrochloride nasal spray 50μg, and placebo nasal spray 50μg
Drug: Placebo — Group 3 (C) was administered 100 μg of placebo nasal spray
  Arms: Group 3(C): Placebo nasal spray 100μg
Drug: Dexmedetomidine hydrochloride nasal spray — Group 2 (HD) was administered 100 μg of dexmedetomidine hydrochloride nasal spray
  Arms: Group 2(HD): Dexmedetomidine hydrochloride nasal spray 100μg

SUMMARY:
The goal of this clinical trial is to assess the viability of dexmedetomidine hydrochloride nasal spray under minimal or no supervision and to further investigate novel clinical applications for this medication. This study aims to investigate the following aspects: the incidence of adverse respiratory and circulatory events requiring medical intervention following the administration of dexmedetomidine nasal spray for pre-anesthetic sedation, its sedative efficacy and onset time, and its impact on the quality of post-anesthesia recovery and the occurrence of postoperative delirium. Researchers will compare dexmedetomidine hydrochloride nasal spray to a placebo (a look-alike substance that contains no drug) to see the incidence and severity of adverse events following administration. Participants will receive either dexmedetomidine nasal spray or a placebo 45 minutes before anesthesia induction. The blinded assessor will continuously monitor and record vital signs, adverse events, and the level of sedation. More importantly, observations and records should be made for respiratory and circulatory events that require medical intervention. A follow-up assessment will be conducted within three days after the operation to evaluate the incidence of postoperative delirium and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older, including the age of 18; no gender limitation;
* American Society of Anesthesiologists (ASA) grade I to III;
* Require general anesthesia, intraspinal anesthesia, or nerve block anesthesia for an elective surgical procedure;
* Provide informed consent for participation in this study prior to the commencement of the trial and execute a written document of informed consent willingly.

Exclusion Criteria:

* Individuals with a known hypersensitivity to dexmedetomidine hydrochloride or any excipient; patients with a documented allergy to any tranquilizers, opioids, or other substances employed in the trial;
* Individuals with airway hyperactivity, such as those suffering from chronic obstructive pulmonary disease (COPD), asthma, or sleep apnea, who are determined by the researchers to have experienced or are experiencing safety concerns related to these conditions;
* Patients with a history of nasal disorders, previous surgical procedures, or allergic reactions deemed clinically significant by the research team, which could significantly impact drug absorption (e.g., chronic nasal congestion, rhinorrhea, nosebleeds, and other symptoms, as well as anatomical or mucosal abnormalities in the nose that may affect drug uptake);
* A blood oxygen saturation (SpO2) level of less than or equal to 92% in a non-oxygenated state during the screening period;
* patients with current psychiatric disorders (like schizophrenia or depression) or cognitive impairment; those with a history of epilepsy; or individuals with a past record of psychotropic or narcotic substance abuse;
* A history of myocardial infarction or unstable angina pectoris within the past six months prior to the screening phase;
* A heart rate or pulse rate of less than or equal to 50 beats per minute during the screening period, the presence of clinically significant heart functional abnormalities as determined by the investigators, or the presence of grade II or higher atrioventricular block (excluding patients with implanted pacemakers) along with other severe arrhythmias;
* Patients with inadequately controlled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg during the screening period) or hypotension (systolic blood pressure ≤90 mmHg and/or diastolic blood pressure ≤ mmHg during the screening period);
* Participants who have already engaged in other clinical trials and have taken the investigational drug within the three months preceding the screening period;
* Pregnant or lactating women expected to undergo a cesarean section during labor and delivery;
* The investigator concludes that the patient possesses other conditions rendering them ineligible for trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events in the circulatory and respiratory system requiring medical intervention | 45 minutes after administration, before the induction of anesthesia

SECONDARY OUTCOMES:
Ramsay score | 45 minutes after administration, before the induction of anesthesia
  The Ramsay Sedation Scale is a widely used tool to assess the level of sedation in patients; a higher level indicates a stronger sedative effect.
  Level 1 : Anxiety, with agitation or restlessness. Level 2 : Calm and cooperative, with orientation to time and place. Level 3 : Responds to commands, but with delayed or slurred speech. Level 4 : Sleepy, but easily arousable to voice. Level 5 : Sleepy, with a slow response to voice. Level 6 : Deeply sedated, with no response to voice or light stimulation.
The time from the end of the surgery to the first postoperative Aldrete score ≥ 9 | Day 1
The incidence of circulatory and respiratory adverse events that require medical intervention as determined by researchers from the end of surgery to the exit of PACU | From the end of surgery to the exit of PACU
Incidence of POD | Within 72 hours after the surgery was completed
Postoperative patient and anesthesiologist satisfaction score | Within 72 hours after the surgery was completed
  The patients and the anesthesiologists rated the satisfaction of this anesthesia on a scale of 1 to 10. The higher the score, the higher the level of satisfaction.

IPD SHARING:
Plan to Share IPD: No